CLINICAL TRIAL: NCT00316459
Title: A Randomized, Double-Blind, Placebo and Moxifloxacin (Open-Label) Controlled, 4-Period, Crossover Study of the Effects of Multiple Oral Doses of ERB-041 on Cardiac Repolarization in Healthy Subjects
Brief Title: Study Evaluating the Effects of Multiple Oral Doses of ERB-041 on Cardiac Repolarization in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A2-110
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Healthy; Long QT Syndrome
Keywords: Healthy; Cardiac; Pharmacokinetics
MeSH Terms: conditions — Long QT Syndrome | interventions — ERB 041

INTERVENTIONS:
Drug: ERB-041

SUMMARY:
To assess the effect of ERB-041 after multiple oral doses on cardiac repolarization as assessed by the QTc interval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and ECG.
* Nonsmoker or smoker of fewer than 10 cigarettes (half a pack) per day as determined by history.

Exclusion Criteria:

* A family history of long QT syndrome and/or cardiac death.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematological, neurological, or psychiatric disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64
Dates: Start 2006-05

PRIMARY OUTCOMES:
To assess the effect of ERB-041 after multiple oral doses on cardiac repolarization as assessed by the QTc interval

SECONDARY OUTCOMES:
To characterize pharmacokinetic and pharmacodynamic relationships as it relates to QTc.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Miami, Florida, United States